CLINICAL TRIAL: NCT06164600
Title: Bovine Colostrum Supplementation for Prophylaxis Against Recurrent Urinary Tract Infection in Children
Brief Title: Bovine Colostrum for Prophylaxis Against Recurrent Urinary Tract Infection in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Usama Hashem, lecturer of Pediatrics, Nephrology Department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMAUS MS 2444/2023
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2023-12

CONDITIONS: Urinary Tract Infections; Recurrent; Child; Prevention & Control; Infections; Urologic Diseases; Communicable Diseases
Keywords: Bovine Colostrum
MeSH Terms: conditions — Urinary Tract Infections; Recurrence; Infections; Urologic Diseases; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovine Colostrum group (Experimental): Thirty Patients will receive oral bovine colostrum sachets daily for one month in a dose of 1 sachet per day for children less than 2 years and 2 sachets per day for children older than 2 years.They will be instructed to take each sachet on an empty stomach at least 30 min before meals after being added to 50 ml of neutral (previously boiled) water with continuous mixing until being dissolved.
  Interventions: Dietary Supplement: Bovine colostrum
- Control group (Placebo Comparator): Thirty Patients will receive oral placebo sachets daily in a similar dose for the same duration. They will be instructed to receive it similarly to the experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Bovine colostrum — A powdered form of the first 6 hours bovine colostrum [65 mg lactoferrin, lactoperoxidase: 2.8 unit and immunoglobulins in the form of 350 mg IgG, 35.3 mg of Ig A and 25.3 mg Ig M]
  Other Names: ImmuGuard®
  Arms: Bovine Colostrum group
Drug: Placebo — Oral placebo sachets will be provided by ImmuGuard® manufacturing company.
  Arms: Control group

SUMMARY:
Prebiotics as bovine colostrum are considered as a valuable supplement in the prevention of upper respiratory tract infections, gastrointestinal tract infections and neonatal sepsis. It contains many bioactive substances, such as immunoglobulins, lactoferrin, lysozyme, lactoperoxidase, and other growth factors.There is a lack of research on the use of prebiotics for prophylaxis against recurrent urinary tract infection (UTI) in children.In this era of increasing bacterial resistance to antimicrobial therapy, bovine colostrum can offer an approach for prophylaxis against UTI in these patients.We aim at this trial to evaluate the efficacy and safety of bovine colostrum as a prebiotic for prophylaxis against recurrent urinary tract infection in children.

DETAILED DESCRIPTION:
This prospective,randomized, placebo-controlled pilot study will enroll a total of sixty children diagnosed with recurrent UTI and following up in Pediatric Nephrology Clinic at Children's Hospital at Ain Shams University. Participants' parents will sign an informed consent statement prior to inclusion in the study. Children fulfilling the eligibility criteria, whether they are already on antibiotic prophylaxis for UTI or not, will be randomly assigned (1:1), using a computer-generated list into one of two groups: Experimental group receiving oral Bovine colostrum sachets daily for 1 month (n=30)& Control group receiving oral placebo sachets daily for the same duration(n=30).

* Patient demographics, clinical symptoms suggestive of UTI, medication history, any risk factors for UTI, and clinical examination will be obtained at baseline.These will be followed up monthly for 6 months after the beginning of the study either during clinic visits or via telephone calls.
* Urine analysis (UA) will be done at base line, and monthly for 6 months. However if symptoms suggestive of UTI, UA will be requested.
* Urine culture at base line and with the appearance of symptoms or presence of pyuria in the urine analysis defined by > 10 WBC /HPF.

ELIGIBILITY:
Inclusion Criteria:

* Documented recurrent UTI proven by positive urine culture. Recurrent UTI will be defined according to NICE guidelines as any of the following:

  1. 2 or more episodes of UTI with acute pyelonephritis.
  2. 1 episode of UTI with acute pyelonephritis plus 1 or more episode of UTI with cystitis.
  3. 3 or more episodes of UTI with cystitis.

Exclusion Criteria:

1. Allergy or hypersensitivity to the prescribed prebiotic.
2. Presence of any endo-urinary device (ureteral stent).
3. Presence of urinary stones

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Number of symptomatic UTIs | 6-months follow-up period.
  defined as the presence of bacteriuria (bacterial colony count ≥100,000 through clean catch method or ≥ 50000 CFU/ml through urinary catheter, IN COMBINATION with the presence of at least 1 acute (<48 hours) clinical sign of infection (fever, shivers, vomiting, loin pain, dysuria, heamturia). Data regarding the type of UTI and the causative organism will be reported.
Number of UTIs with urinary bacterial colony count through urinary catheter > 10,000 CFU/ml having fever and pyuria | 6-months follow-up period.
  European guidelines state that growth of 10,000 CFU/mL or even 1,000 CFU/ml are sufficient to diagnose a UTI from a catheterized urine while US and Canadian guidelines use 50,000 CFU/mL as the cut-off

SECONDARY OUTCOMES:
Number of patients with asymptomatic bacteruria | 6-months follow-up period.
  defined as asymptomatic patients having bacterial colony count :
  * 100,000 CFU/ml through clean catch method OR
  * 50,000 CFU/ml through urinary catheter
Number of asymptomatic patients with bacterial colony count > 10.000 CFU/ml and< 50,000 for specimen collected by urinary catheter. | 6-months follow-up period.
  Since the strict definition of bacterial colony count in UTI is operational and not absolute, the Italian Society of Pediatric nephrology issued guidelines recommended the threshold for specimen collected by catheterization to be >50.000 CFU/mL5, Or >10.000 CFU/mL if fever and leucocyturia are present.
Number of symptomatic infections elsewhere GIT/respiratory | 6-months follow-up period.
Adverse effects to the prescribed bovine colostrum: GIT problems or allergy | 6-months follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Pediatric Hospital, Cairo, Abbasseiya, Egypt

REFERENCES:
- [Background] Ammenti A, Alberici I, Brugnara M, Chimenz R, Guarino S, La Manna A, La Scola C, Maringhini S, Marra G, Materassi M, Morello W, Nicolini G, Pennesi M, Pisanello L, Pugliese F, Scozzola F, Sica F, Toffolo A, Montini G; Italian Society of Pediatric Nephrology. Updated Italian recommendations for the diagnosis, treatment and follow-up of the first febrile urinary tract infection in young children. Acta Paediatr. 2020 Feb;109(2):236-247. doi: 10.1111/apa.14988. Epub 2019 Oct 6. PMID 31454101
- [Background] Ammenti A, Cataldi L, Chimenz R, Fanos V, La Manna A, Marra G, Materassi M, Pecile P, Pennesi M, Pisanello L, Sica F, Toffolo A, Montini G; Italian Society of Pediatric Nephrology. Febrile urinary tract infections in young children: recommendations for the diagnosis, treatment and follow-up. Acta Paediatr. 2012 May;101(5):451-7. doi: 10.1111/j.1651-2227.2011.02549.x. Epub 2012 Jan 3. PMID 22122295
- [Background] Robinson JL, Finlay JC, Lang ME, Bortolussi R; Canadian Paediatric Society, Infectious Diseases and Immunization Committee, Community Paediatrics Committee. Urinary tract infections in infants and children: Diagnosis and management. Paediatr Child Health. 2014 Jun;19(6):315-25. doi: 10.1093/pch/19.6.315. PMID 25332662
- [Background] Stein R, Dogan HS, Hoebeke P, Kocvara R, Nijman RJ, Radmayr C, Tekgul S; European Association of Urology; European Society for Pediatric Urology. Urinary tract infections in children: EAU/ESPU guidelines. Eur Urol. 2015 Mar;67(3):546-58. doi: 10.1016/j.eururo.2014.11.007. Epub 2014 Dec 2. PMID 25477258
- See also: Related Info — https://www.nice.org.uk/guidance/ng112